CLINICAL TRIAL: NCT01693848
Title: Molecularly Imprinted Polymer Sensors of Modified Nucleosides for Non-invasive Monitoring, of Cancer Therapy: Impact of Surgical Resection of Metastasis on Urinary Excretion of Modified Nucleosides.
Brief Title: "Cancersensor" Metastasis Resection
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C11-58; 2012-A00011-42 (Registry Identifier: IDRCB)
Record Dates: First submitted 2012-09-07; First posted 2012-09-26 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Colorectal; Cancer; Metastatic; Control; Urine; Nucleosides; Surgery; General anesthesia; Scheduled for surgery
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients: Patients with metastatic colorectal cancer scheduled for metastatic surgery
- Control patients: Patients with metastatic colorectal cancer scheduled for general anesthesia without metastatic surgery

SUMMARY:
Observational, non randomized study aimed at measuring the effect of surgical resection of metastasis in the urinary concentrations of physiological modified nucleosides in 45 patients with metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed metastatic colorectal cancer;
* 0 to 3 prior chemotherapy lines; Signed informed consent;
* Good understanding of the protocol and of the follow-up;
* Estimated life expectancy exceeding 3 months;
* At least one measurable metastatic lesion (RECIST criteria);
* Performance Status (WHO) of 0 to 2;
* Good haematological, hepatic and renal functions.

Exclusion Criteria:

* Poor haematological, hepatic or renal functions;
* Uncontrolled chronic disease;
* Serious unhealed wound, ulcer or fracture within the previous month;
* Clinical or laboratory finding suggesting possible abnormalities in nucleosides urinary excretion;
* Pregnancy or breast-feeding during the previous month;
* Transmeridian trip of more than 4 time zones within the prior 2 weeks;
* Person with legal restriction to participate into clinical research, according to the current law in France.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic colorectal cancer treated at the Department of Medical Oncology of Paul Brousse Hospital
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2012-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Effect of resection of metastasis on urinary excretion of modified nucleosides | 10 days
  1 Urine sample per day 3 before and 7 after surgery Measurement of modified nucleoside concentration

SECONDARY OUTCOMES:
Identification of modified nucleosides as biomarkers for colorectal cancer | 10 days
  Measurement of modified nucleosides in urine samples before and after metastatic resection

CONTACTS AND LOCATIONS:
Locations (1):
- Paul Brousse hospital, Villejuif, France